CLINICAL TRIAL: NCT03059498
Title: Determining Plasma Bupivacaine Levels Following Pectoral Nerve Blocks: A Prospective Observational Study
Brief Title: PECS Block: Plasma Bupivacaine Level
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00042325
Record Dates: First submitted 2017-02-14; First posted 2017-02-23 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Nerve Blocks
Keywords: PECS I and II; PECS blocks
MeSH Terms: interventions — Dental Occlusion; Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- unilateral PECS block patients (Active Comparator): unilateral PECS I and II block using bupivacaine
  Interventions: Procedure: Unilateral PECS I and II block; Drug: Bupivacaine
- bilateral PECS block patients (Active Comparator): bilateral PECS I and II block using bupivacaine
  Interventions: Procedure: Bilateral PECS I and II block; Drug: Bupivacaine

INTERVENTIONS:
Procedure: Unilateral PECS I and II block — A truncal block called the pectoralis nerve block (PECS I and II block). Unilateral. Using Bupivacaine
  Arms: unilateral PECS block patients
Procedure: Bilateral PECS I and II block — A truncal block called the pectoralis nerve block (PECS I and II block). Bilateral. Using Bupivacaine.
  Arms: bilateral PECS block patients
Drug: Bupivacaine — Bupivacaine solution 0.25%. At the PECS I site each patient will receive 10 cc of local anesthetic solution, and at the PECS II site an additional 20 cc of local anesthetic solution will be placed.

SUMMARY:
The purpose of this study is to determine peak plasma bupivacaine concentrations in a similar fashion for PECS I/II blocks. The investigators hypothesis is that the mean peak plasma levels for patients undergoing PECS I/II blocks will be less than the levels reported to cause early neurotoxicity of [2.2 (0.9) micrograms/ml]6 in patients receiving intravenous bupivacaine infusions.

DETAILED DESCRIPTION:
Regional anesthesia techniques are common modalities used to provide analgesia following both upper and lower extremity surgeries. It is also often used for truncal procedures for the same purpose. A relatively new truncal block, first described in 2012 by Blanco, called the pectoralis nerve block (PECS I and II block) has been used successfully for breast surgery1-3. Despite its description and success in clinical practice, the extent of systemic absorption from this truncal plane block has not been described to date. However, in a study published in the British Journal of Anesthesia, this has been done for another truncal plane block, the transverse abdominus plane (TAP) block where the local anesthetic was noted to peak and had a mean total concentration of ropivacaine occurring at 30 minutes after the block4. During this study, samples were taken at 10, 20, 30, 45, 60, 90, 120, 180, and 240 minutes. The investigators anticipate that since this is a similar truncal plane block, absorption will be comparable in terms of timing. However, the concentration of drug absorbed may be different given the proximity to the ribs, intercostal and thoracic vasculature, and a higher concentration of local given the smaller plane for local anesthetic spread. Given that the investigators want to find the peak of the curve and the peak concentration of bupivacaine from the PECS block, the investigators feel will need 5 samples at the times outlined below. This number of samples was chosen to approximate a study published in 2004 where ten subjects received ropivacaine for scalp blocks and serum ropivacaine levels were measured at 15, 30, 45, 60, 90, and 120 minutes5. The investigators feel that the 120 minute measurement is well beyond the peak plasma level of bupivacaine given the findings in the TAP and scalp studies. Therefore,the investigators will collect the following samples at these times after the block is completed: 5, 10, 20, 40, 60, and 90 minutes. The purpose of this study is to determine peak plasma bupivacaine concentrations in a similar fashion for PECS I/II blocks. The investigators hypothesis is that the mean peak plasma levels for our patients undergoing PECS I/II blocks will be less than the levels reported to cause early neurotoxicity of [2.2 (0.9) micrograms/ml]6 in patients receiving intravenous bupivacaine infusions.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving a unilateral PECS I and II block for any surgery being provided by Wake Forest Baptist Medical Center

Exclusion Criteria:

* Subjects with contraindications to regional anesthesia, such as a history of allergy to amide local anesthetics,
* presence of a progressive neurological deficit,
* a pre-existing coagulopathy,
* infection at site of injection.
* or the following conditions:
* patient receiving any other additional local anesthetic from another procedure
* infection over site of block
* patient refusal
* significant renal or liver dysfunction on laboratory analysis
* weight <60 kg
* pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2017-11-15 (Actual)

PRIMARY OUTCOMES:
Peak plasma bupivacaine concentration | 90 minutes after dose
  Will be determined by samples collected at these times after the block is completed: 5, 10, 20, 40, 60, and 90 minutes
Bupivacaine mean concentration | 90 Minutes after dose
  Calculated from samples at these times after the block is completed: 5, 10, 20, 40, 60, and 90 minutes
Standard deviations of plasma bupivacaine concentrations | 90 minutes after dose
  Will be calculated using samples at these times after the block is completed: 5, 10, 20, 40, 60, and 90 minutes

SECONDARY OUTCOMES:
Rates of block success | 30 minutes after block
  As assessed by pin prick at the mid-clavicular line overlying the pectoralis major in between the dermatomes of T2 to T4.
Rates of adequate ultrasound success of appropriate separation of the muscular layers for each block. | At the end of the block placement, 0 minutes timepoint.
  be rated clinically on a 3 point scale: 0 = very poor spread with possible block failure, 1 = initially poor spread, but layers separated appropriately with high chance for successful block, 2 = spread clearly seen to separate muscular layers and successful block anticipated.
Rates of symptoms of local anesthetic systemic toxicity | 90 minutes after block
  Presence of symptoms from the end of the block to 90 minutes after the block.

CONTACTS AND LOCATIONS:
Overall Officials: J. Douglas Jaffe, DO, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No